CLINICAL TRIAL: NCT02470702
Title: A Double-Blind Randomized Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple 1200 mg Dose Intravenous Oritavancin Infusions in Healthy Subjects
Brief Title: Multiple Oritavancin Doses on Safety, Tolerability, and Pharmacokinetics in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MDCO-ORI-15-02
Record Dates: First submitted 2015-05-08; First posted 2015-06-12 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — oritavancin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oritavancin (Experimental): Subjects randomized to oritavancin will receive four doses (Cohort 1) or eight doses (Cohort 2) of 1200 mg oritavancin, infused intravenously over 3 hours
  Interventions: Drug: Oritavancin
- Placebo (Placebo Comparator): Subjects randomized to placebo will receive four doses (Cohort 1) or eight doses (Cohort 2) of 1000 mL D5W, infused intravenously over 3 hours
  Interventions: Drug: Placebo (D5W)

INTERVENTIONS:
Drug: Oritavancin
  Arms: Oritavancin
Drug: Placebo (D5W)
  Arms: Placebo

SUMMARY:
This protocol describes a double-blind study to evaluate the safety and pharmacokinetics of multiple IV doses of 1200 mg ORBACTIV (oritavancin) in healthy subjects.

DETAILED DESCRIPTION:
Oritavancin has been approved in the United States for the treatment of adult patients with acute bacterial skin and skin structure infections (ABSSSIs) caused or suspected to be caused by susceptible isolates of designated Gram-positive microorganisms. The purpose of this study is to determine the (a) safety and tolerability and (b) pharmacokinetic profile of multiple doses of Oritavancin given over a 7-8 week period.

Cohort 1 will consist of 14 subjects, randomized to receive a total of four doses of either oritavancin or placebo, given once every two weeks in a double-blind fashion.

After completion of cohort 1, a Data Safety Monitoring Board will review the blinded safety data and pharmacokinetics (PK) for cohort 1 and determine whether to continue with cohort 2, modify cohort 2 or end the study. The cohorts for this study are sequential.

Cohort 2 will consist of 14 subjects, randomized to receive a total of eight doses of either oritavancin or placebo (4 subjects) given once every week in a double-blind fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide written informed consent before initiation of any study-related procedures.
2. Healthy male or female between the ages of 18 and 55 years, inclusive.
3. Body mass index (BMI) < 45 kg/m^2.
4. Subject is in good health based on medical history and physical examination findings and has no clinically meaningful safety laboratory abnormalities (CBC, blood chemistry, and urinalysis) or 12 lead ECG results, as assessed by the PI.
5. Vital signs (BP, pulse and temperature) measured at screening/baseline must be within the following ranges: SBP ≥90 to ≤150 mm Hg, DBP ≥45 to ≤90 mm Hg; Heart Rate ≥ 40 to ≤90 bpm (taken after resting in a supine position for at least 5 minutes).
6. Willing to avoid all medications (other than the study drug and acetaminophen/paracetamol for minor aches/pains) during the study. This includes prescription and non-prescription medications, vitamins, herbal supplements, and nutraceuticals.
7. Subject is a non-smoker and is willing to abstain from alcohol/illegal drug use for the duration of the study.
8. If the female subject is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use at least 2 highly effective methods of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, abstinence) or male partner sterilization alone for the duration of the study until 60 days after study drug administration.

Exclusion Criteria:

1. Has any condition, including findings in the medical history or in pre-study assessments that constitutes a risk or a contraindication for the participation in the study or completing the study.
2. Female subjects of childbearing potential that have a positive test result for human chorionic gonadotropin (hCG) at screening.
3. Female subjects who are nursing.
4. Positive urine test for alcohol and/or for drugs of abuse at screening.
5. Has a history or presence of alcohol/drug abuse within 2 years. Alcohol abuse is defined as regularly consuming >3 units/day (21 units per week for men), >2 units/day (14 units/week) for women. 1 unit of alcohol is defined as a can of 4% beer (330 mL), approximately 190 mL of 6-7% beer (malt liquor), a glass of 40% spirits (30 mL), or a glass of wine (100 mL).
6. History of hypersensitivity to drugs with a similar chemical structure (i.e. glycopeptide antibiotics) to oritavancin or any of its excipients.
7. Blood or plasma donation within the past 2 months.
8. Subjects who participated in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days or 5 half-lives, whichever is longer, prior to screening and/or unwilling to allow at least two months before participation in another drug trial following the current trial.
9. Treatment with any prescription or OTC drugs, within 2 weeks or 5 half-lives, whichever is longer, or herbal nutritional supplements within 2 weeks of screening, with the exception of acetaminophen/paracetamol for minor aches/pains. Subjects will not be allowed to receive medications for the duration of the study (except the above-mentioned acetaminophen/paracetamol). Birth control or other hormone replacement is also permitted as long as it has been taken at a stable dose for at least three months before the screening visit and remains stable for the duration of the study.
10. Males who are unwilling to practice abstinence or use an acceptable method of birth control during the entire study period (i.e. condom with spermicide).
11. Subjects that have any surgical or medical condition that could interfere with the administration of the study drug.
12. Subjects that have known active hepatitis B or C, or human immunodeficiency virus (HIV) infection or has known immune deficiency disease at screening.
13. Subjects that have any condition that would confound or interfere with the assessment of safety.
14. Subjects that have poor IV access as determined by the investigator. Subjects excluded for any of the previous criteria may only be rescreened for participation after discussion with sponsor and principal investigator.
15. Prior exposure to Oritavancin alone or in combination with another product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability: AEs/SAEs | From consent until day 110 safety follow up call
  a composite measure of the number and types of AEs/SAEs encountered and relationship to time of dosing
Safety & Tolerability: clinical safety laboratory results | From consent until day 110 safety follow up call
  A composite measure of multiple laboratory results assessing the clinical significance of any changes from baseline
Safety & Tolerability: vital sign measurements | From consent until day 110 safety follow up call
  A composite of multiple vital sign measurements, assessing the clinical significance of any changes from baseline
Safety & Tolerability: ECGs | From consent until day 110 safety follow up call
  A composite of multiple ECG measurements, assessing the clinical significance of any changes from baseline
Safety & Tolerability: physical examination findings | From consent until day 110 safety follow up call
  A composite of multiple physical examination findings, assessing the clinical significance of any changes from baseline

SECONDARY OUTCOMES:
Pharmacokinetics: AUC0-last | From pre-dose until 720 hours past last dose
  AUC from time zero to the time of the last measurable concentration
Pharmacokinetics: AUC0-72 | From pre-dose until 72 hours past last dose
  AUC from time zero to 72 hours post dose
Pharmacokinetics: AUC0-∞ | From pre-dose until 720 hours past last dose
  AUC from time zero to infinity
Pharmacokinetics: Cmax | From pre-dose until 720 hours past last dose
  maximum measured plasma concentration
Pharmacokinetics: Cmin | From pre-dose until 720 hours past last dose
  minimum plasma concentration
Pharmacokinetics: Tmax | From pre-dose until 720 hours past last dose
  time to Cmax
Pharmacokinetics: t1/2 | From pre-dose until 720 hours past last dose
  elimination half- life
Pharmacokinetics: CL | From pre-dose until 720 hours past last dose
  total body clearance
Pharmacokinetics: VSS | From pre-dose until 720 hours past last dose
  Volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- West Bend, Wisconsin, United States